CLINICAL TRIAL: NCT02968433
Title: The Stanford Parkinson's Disease Plasma (SPDP) Study: Intravenously-Administered Plasma From Young Donors for Treatment of Moderate Parkinson's Disease
Brief Title: The Stanford Parkinson's Disease Plasma Study
Acronym: SPDP
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Helen M. Bronte-Stewart, Primary Investigator, Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB 38417
Record Dates: First submitted 2016-11-14; First posted 2016-11-18 (Estimated); Results first posted 2020-12-30 (Actual); Last update posted 2020-12-30 (Actual); Status verified 2020-12

CONDITIONS: Parkinson Disease(PD)
Keywords: Young Male Plasma
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Infusions of Young Plasma (Experimental): All participants will undergo neuropsychological, neuropsychiatric, and kinematic assessments prior to receiving infusions of young plasma as the treatment.
  Participants will receive 1 unit of young plasma, twice a week over a four week duration.
  After the four weeks of plasma infusions, participants will undergo neuropsychological, neuropsychiatric and kinematic reassessments. No deception will be used.
  Interventions: Drug: Infusions of young plasma

INTERVENTIONS:
Drug: Infusions of young plasma — Participants will receive four twice- weekly infusions of 1 unit young plasma (male, ages between 18-25)

SUMMARY:
The purpose of this study is to demonstrate that young plasma infusions can be performed safely in patients with Parkinson's Disease (PD). Secondary outcomes will include behavioral and laboratory data that will support the next study that will inquire whether young plasma infusions improve or slow the progression of cognitive, mood and/or motor impairment and rate markers of the disease.

DETAILED DESCRIPTION:
Parkinson's disease (PD) is a neurodegenerative disease that affects over 1.6 million people in the United States and whose incidence increases with age, affecting over 1% of people over the age of 65. The neuropathological processes involved in PD are widespread throughout the brain, and are reflected in a constellation of motor, cognitive, mood and other non-motor symptoms. Treatments to date have largely focused on dopamine replacement strategies or deep brain stimulation, both symptomatic treatments.

As neurodegenerative diseases progress, there are major changes throughout the body and brain. These changes are transmitted in the body via the circulatory system between organs, tissues and cells. Recent findings from multiple laboratories have shown that infusions of young plasma into aging rodents can have beneficial effects on cognitive functions. This suggests that the circulating components of plasma can improve cognitive and disease-relevant symptoms. This has motivated the field to treat multiple disorders with blood products and their constituent active components.

The established safety of blood transfusions allows the investigators to test whether infusions of young plasma can ease the neurological symptoms in human subjects with neurodegenerative diseases. A related study of plasma infusions has already been completed at Stanford in patients with Alzheimer's disease (ClinicalTrials.gov identifier NCT02256306).

The investigator proposes to test the safety and efficacy of transfusing young plasma into PD participants, in order to establish its effects on motor and cognitive functions in participants in a Phase 1 study. The successful completion of this study will inform the design of future, larger and multicenter studies with the goal to determine whether infusions of young plasma can ameliorate the neurodegenerative symptoms and underlying pathophysiology in Parkinson's disease.

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis of clinically probable or established Parkinson's Disease (MDS criteria)
* Subject must be on a stable dose of dopaminergic medication and/or Deep Brain Stimulation (DBS) parameters for at least 4 weeks prior to screening and for the duration of the study
* Subject must be competent to sign consent
* Subject must be willing to commit to being available for testing and infusions for 6 consecutive weeks (2 testing consecutive weeks, 4 infusion consecutive weeks) followed by two visits a month after final infusion.
* The availability of a study partner who knows the patient well and is willing to accompany the subject to all trial (optional if participant is able to consent and travel by self)

Exclusion Criteria:

* The participation in any other interventional clinical trial
* The inability to travel to Stanford
* Inability to walk without assistance in the off or on medication state
* The clinically determined presence of dementia
* A clinical suspicion/diagnosis of Multiple System Atrophy (MSA), Progressive Supranuclear Palsy (PSP), Lewy Body Dementia (LBD), Essential Tremor (ET)
* Subject's pregnancy or likelihood of pregnancy within the next 6 months.
* Subject's positive test results for Hepatitis B, Hepatitis C or HIV at screening
* Any other condition or situation that the investigator believes may interfere with the safety of the subject or the intent and conduct of the study
* Subject's medical history of:

Stroke Anaphylaxis Gout- may cause an increase in uric acid Prior adverse reaction to any human blood product Any history of a blood coagulation disorder or hypercoagulability Congestive heart failure Uncontrolled hypertension Renal failure Prior intolerance to intravenous fluids Recent history of uncontrolled atrial fibrillation immunoglobulin A deficiency (by history)

* Subject's relation to medications or other treatments:
* Any concurrent use of an anticoagulant therapy. Antiplatelet drugs (e.g., aspirin or clopidogrel) are acceptable.
* The use of Inosine, which may alter urate levels
* Initiation or change in the dosage of a cholinesterase inhibitor or memantine during the trial. A participant already on a cholinesterase inhibitor or memantine must be on a stable dose for at least one month prior to Screening.
* Concurrent participation in another interventional treatment trial for Parkinson's disease. If there was prior participation, the last dose of the investigational agent must have been at least 6 months prior to Screening.
* Treatment with any human blood product, including intravenous immunoglobulin, during the 6 months prior to Screening or during the trial.
* Concurrent daily treatment with benzodiazepines, typical or atypical antipsychotics, long-acting opioids, or other medications that, in the investigator's opinion, interfere with cognition. Intermittent treatment with short-acting benzodiazepines or atypical antipsychotics may be permitted, provided that no dose is administered within the 72 hours preceding any cognitive assessment.

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2019-12 (Actual); Study Completion 2019-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Helen Bronte-Stewart, MS, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford Movement Disorders Clinic, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sha SJ, Deutsch GK, Tian L, Richardson K, Coburn M, Gaudioso JL, Marcal T, Solomon E, Boumis A, Bet A, Mennes M, van Oort E, Beckmann CF, Braithwaite SP, Jackson S, Nikolich K, Stephens D, Kerchner GA, Wyss-Coray T. Safety, Tolerability, and Feasibility of Young Plasma Infusion in the Plasma for Alzheimer Symptom Amelioration Study: A Randomized Clinical Trial. JAMA Neurol. 2019 Jan 1;76(1):35-40. doi: 10.1001/jamaneurol.2018.3288. PMID 30383097
- [Background] Villeda SA, Luo J, Mosher KI, Zou B, Britschgi M, Bieri G, Stan TM, Fainberg N, Ding Z, Eggel A, Lucin KM, Czirr E, Park JS, Couillard-Despres S, Aigner L, Li G, Peskind ER, Kaye JA, Quinn JF, Galasko DR, Xie XS, Rando TA, Wyss-Coray T. The ageing systemic milieu negatively regulates neurogenesis and cognitive function. Nature. 2011 Aug 31;477(7362):90-4. doi: 10.1038/nature10357. PMID 21886162
- [Background] Villeda SA, Plambeck KE, Middeldorp J, Castellano JM, Mosher KI, Luo J, Smith LK, Bieri G, Lin K, Berdnik D, Wabl R, Udeochu J, Wheatley EG, Zou B, Simmons DA, Xie XS, Longo FM, Wyss-Coray T. Young blood reverses age-related impairments in cognitive function and synaptic plasticity in mice. Nat Med. 2014 Jun;20(6):659-63. doi: 10.1038/nm.3569. Epub 2014 May 4. PMID 24793238
- [Result] Parker JE, Martinez A, Deutsch GK, Prabhakar V, Lising M, Kapphahn KI, Anidi CM, Neuville R, Coburn M, Shah N, Bronte-Stewart HM. Safety of Plasma Infusions in Parkinson's Disease. Mov Disord. 2020 Nov;35(11):1905-1913. doi: 10.1002/mds.28198. Epub 2020 Jul 7. PMID 32633860

RESULTS

PARTICIPANT FLOW:
Groups:
- Infusions of Young Plasma: All participants will undergo neuropsychological, neuropsychiatric, and kinematic assessments prior to receiving infusions of young plasma as the treatment.
  Participants will receive 1 unit of young plasma, twice a week over a four week duration.
  After the four weeks of plasma infusions, participants will undergo neuropsychological, neuropsychiatric and kinematic reassessments. No deception will be used.
  Infusions of young plasma: Participants will receive four twice- weekly infusions of 1 unit young plasma (male, ages between 18-25)
Period: Overall Study
Arm/Group | Infusions of Young Plasma
Started | 16
Completed | 15
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Population: Participants who completed the study
Arm/Group | Infusions of Young Plasma
Number analyzed (Participants) | 15
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 8
  >=65 years | 7
Age, Continuous [Mean (Standard Deviation); unit: years] | 63 (8.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 10
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 12
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 15

OUTCOME MEASURES:

1. Primary Outcome: Number of Related and Unrelated Adverse Events
Description: The primary outcome measure is the number of adverse events across all participants that might be related to young plasma infusions as a novel treatment to Parkinson's Disease symptoms. Adverse events were categorized as probably, possibly, or not related to the study intervention.
Time Frame: 8 weeks
Measure: Number; unit: events
Arm/Group | Infusions of Young Plasma
Number analyzed (Participants) | 16
events
  Number of probably related AEs | 14
  Number of possibly related AEs | 3
  Number of unrelated AEs | 36

2. Other Pre Specified Outcome: Change in Quantitative Data of Cognitive Ability (Neuropsychological Battery)
Description: Change in quantitative data of cognitive ability. Raw scores and normative scores were calculated for all measures according to standardized procedures across all 3 time points.
  The cognitive test battery included:
  * Trail Making Test Part A (0-92; lower scores indicate better performance) and B (0-300; lower scores indicate better performance)
  * Digit Symbol Modalities Test (Oral: 0-110 and Written: 0-110; higher scores indicate better performance)
  * Animal Naming Test (0-no maximum; higher scores indicate better performance)
  * Controlled Oral Word Association Test (COWAT) (0-no maximum; higher score indicates better performance)
  * CogStateTM Groton Maze Learning Test (GML) (minimum score is 0; lower scores indicate better performance)
  * Wechsler Abbreviated Scale of Intelligence-II (WASI-II) Block Design (0-71; higher scores indicate better performance) and Matrix Reasoning (0-30; higher scores indicate better performance)
Time Frame: 8 weeks
Population: Participants who completed the protocol are included in the analysis.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Groups:
- Baseline: Before any treatment-related intervention began
- Immediate-post Evaluation: Immediately after the last plasma infusion
- Delayed-post Evaluation: 4-weeks after the last plasma infusion
Arm/Group | Baseline | Immediate-post Evaluation | Delayed-post Evaluation
Number analyzed (Participants) | 15 | 15 | 15
score on a scale
  WASI-II Block Construction | 34.73 [27.45 to 42.02] | 35.60 [28.32 to 42.88] | 37.47 [30.18 to 44.75]
  WASI-II Matrix Reasoning | 17.47 [14.87 to 20.06] | 17.27 [14.67 to 19.86] | 20.13 [17.54 to 22.73]
  Symbol Digit Modalities Test - Written | 44.80 [39.14 to 50.46] | 47.07 [41.40 to 52.73] | 49.40 [43.74 to 55.06]
  Symbol Digit Modalities Test - Oral | 53.67 [46.89 to 60.44] | 57.40 [50.62 to 64.18] | 57.73 [50.96 to 64.51]
  Trail Making Test-A | 32.53 [27.63 to 37.44] | 29.27 [24.36 to 34.17] | 29.07 [24.16 to 33.97]
  Trail Making Test-B | 83.20 [62.64 to 103.76] | 72.87 [52.31 to 93.42] | 73.53 [52.98 to 94.09]
  Phonemic fluency (COWAT; Letters-FAS) | 43.13 [34.75 to 47.52] | 44.73 [38.35 to 51.12] | 48.07 [41.68 to 54.45]
  Semantic fluency (Animal naming) | 21.40 [19.17 to 23.63] | 22.40 [20.17 to 24.63] | 23.07 [20.84 to 25.29]
  CogState (GML) | 71.47 [53.15 to 89.79] | 54.87 [36.55 to 73.19] | 60.53 [42.21 to 78.85]

3. Other Pre Specified Outcome: Change in Quality of Life
Description: Quality of life (QOL) changes were tracked using the self-report Parkinson's Disease Questionnaire-39 (PDQ-39). The PDQ-39 includes 8 sub-scales: Mobility (raw score range 0-40), Activities of Daily Living (raw score range 0-24), Emotional Well-Being (raw score range 0-24), Stigma (raw score range 0-16), Social Support (raw score range 0-12), Cognition (raw score range 0-16), Communication (raw score range 0-12), and Bodily Discomfort (raw score range 0-12). Subscales scores are totaled then converted to a percentage to calculate the Total score (0 to 100, higher scores indicating the more problems). Ratings are based on participant experiences over the course of the prior month. Lower scores represent better quality of life for all scores.
Time Frame: 8 weeks
Population: Participants who completed the protocol are included in the analysis.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Baseline | Immediate-post Evaluation | Delayed-post Evaluation
Number analyzed (Participants) | 15 | 15 | 15
score on a scale
  Total PDQ-39 Score | 71.81 [59.51 to 84.10] | 66.73 [54.49 to 78.98] | 64.40 [52.16 to 76.64]
  Mobility | 17.33 [13.38 to 21.28] | 16.47 [12.53 to 20.41] | 15.80 [11.86 to 19.74]
  Activities of Daily Living | 12.05 [10.29 to 13.82] | 11.60 [9.85 to 13.35] | 10.53 [8.79 to 12.28]
  Emotional Well-Being | 10.60 [7.75 to 13.45] | 10.13 [7.30 to 12.97] | 10.00 [7.16 to 12.84]
  Stigma | 7.42 [6.22 to 8.63] | 6.20 [5.01 to 7.39] | 5.53 [4.34 to 6.72]
  Social support | 5.57 [3.99 to 7.16] | 5.00 [3.43 to 6.57] | 5.33 [3.76 to 6.90]
  Cognition | 6.90 [5.53 to 8.28] | 6.87 [5.50 to 8.23] | 6.80 [5.43 to 8.17]
  Communication | 5.33 [4.31 to 6.36] | 5.20 [4.19 to 6.21] | 4.60 [3.59 to 5.61]
  Bodily Discomfort | 6.53 [5.25 to 7.82] | 5.27 [4.00 to 6.53] | 5.80 [4.53 to 7.07]

4. Other Pre Specified Outcome: Change in Quantitative Data of Motor Movements up to 8 Weeks
Description: The second outcome measure is the change in the quantitative data of current motor movement ability.
  Patients completed a repetitive Wrist Flexion Extension (rWFE) task with both hands, off therapy at the baseline, immediate-post, and delayed-post visits. Patients were instructed to flex and extend their hands at the wrist as quickly as possible after a "Go" command was given and to stop when instructed. This movement was self-paced, lasted 30 seconds, and was measured using wearable sensors attached to the dorsum of each hand (Motus Bioengineering, Inc.). Variables of interest included the mean angular velocity (Vrms), the variability of mean angular velocity, (CV Vrms), and rhythmicity, defined as the regularity of the interstrike interval (CV ISI). MA = more affected; LA = less affected.
Time Frame: 8 weeks
Population: Patients who completed the rWFE task at baseline and at both outcome visits and who had analyzable data are included in the analysis.
Measure: Mean (95% Confidence Interval); unit: Degrees/sec
Groups:
- Baseline: Baseline rWFE task was completed before any treatment-related intervention.
- Immediate-post Evaluation: Immediate-post rWFE task was completed on the day following the last infusion.
- Delayed-post Evaluation: Delayed-post rWFE task was completed 4-weeks after the final infusion.
Arm/Group | Baseline | Immediate-post Evaluation | Delayed-post Evaluation
Number analyzed (Participants) | 12 | 12 | 12
Degrees/sec
  MA Vrms | 305.13 [196.72 to 413.54] | 339.66 [231.24 to 448.07] | 312.39 [203.98 to 420.81]
  MA CV Vrms | 0.29 [0.2 to 0.38] | 0.19 [0.10 to 0.29] | 0.26 [0.17 to 0.35]
  MA CV ISI | 0.16 [0.07 to 0.26] | 0.11 [0.01 to 0.20] | 0.17 [0.08 to 0.27]
  LA Vrms | 414.47 [295.08 to 533.86] | 411.26 [291.87 to 530.65] | 403.00 [283.61 to 522.39]
  LA CV Vrms | 0.16 [0.09 to 0.22] | 0.17 [0.12 to 0.24] | 0.18 [0.11 to 0.24]
  LA CV ISI | 0.09 [0.05 to 0.14] | 0.09 [0.04 to 0.13] | 0.10 [0.05 to 0.15]

ADVERSE EVENTS:
Time Frame: Adverse events were monitored during the entirety of the trial, starting at baseline and continuing through the 4 week post-infusion mark (8 week total).
Description: Adverse events were categorized using the CTCAE v4.0.
Arm/Group | Infusions of Young Plasma
All-Cause Mortality (participants affected / at risk) | 0/16
Serious Adverse Events (participants affected / at risk) | 0/16
Other Adverse Events (participants affected / at risk) | 13/16
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Infusions of Young Plasma (N=16)
Bruising (Skin and subcutaneous tissue disorders) | 1 (1)
Skin and subcutaneous tissue disorder (Skin and subcutaneous tissue disorders) | 8 (15)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Hypotension (Blood and lymphatic system disorders) | 1 (1)
Nervous system disturbance (Nervous system disorders) | 3 (4)
Bloating (Gastrointestinal disorders) | 1 (1)
Urinary frequency distrubance (Renal and urinary disorders) | 2 (2)
Stomach pain (Gastrointestinal disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Musculoskeletal and connective tissue disorder (Musculoskeletal and connective tissue disorders) | 3 (4)
Chest tightness (General disorders) | 1 (1)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Fall (General disorders) | 1 (1)
Flu-like symptoms (General disorders) | 2 (2)
Tremor (General disorders) | 1 (1)
Involuntary movement (General disorders) | 5 (8)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Sleep disturbance (General disorders) | 2 (2)
Headache (General disorders) | 2 (2)
Gastrointestinal disorders (Gastrointestinal disorders) | 1 (1)
Pain in extremity (General disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-07-23): https://cdn.clinicaltrials.gov/large-docs/33/NCT02968433/Prot_SAP_000.pdf